CLINICAL TRIAL: NCT06334575
Title: Molecular Signatures Associated With Response to ICS Treatment in Patients With COPD Stratified by Eosinophil Levels
Acronym: 3TR-ICS-COPD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Maria Joyera Rodríguez (Other)
Responsible Party: Sponsor-Investigator, Maria Joyera Rodríguez, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-505245-13-00
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICS treatment (Active Comparator)
  Interventions: Drug: Budesonide
- No ICS treatment (No Intervention)

INTERVENTIONS:
Drug: Budesonide — receive, on top of their usual treatment Budesonide dry powder inhaler, 400 mcg/12 hours for 8 weeks
  Arms: ICS treatment

SUMMARY:
The 3TR-ICS COPD study is an international, multicentre, randomized, parallel, controlled study that will recruit clinically stable former smokers COPD patients (with no exacerbations in the previous 8 weeks) on treatment with dual long-acting bronchodilators (LABA+LAMA), minimum 8 weeks of usage, not receiving ICS (either naïve or > 3 months since last usage). The overall objective of this clinical trial is to identify the molecular signatures associated with the molecular response to ICS treatment in patients with COPD stratified by the levels of circulating eosinophils, and the potential influence of the pulmonary microbiome

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥40 years of age.
* ≥ 10 pack-years smoking.
* Former smokers (≥6 months).
* post-bronchodilator FEV1/FVC<0.70.
* FEV1 ≥30 <80% ref.
* Signed written informed consent form.
* On regular treatment with dual long-acting bronchodilators (LABA+LAMA), minimum 8 weeks of usage.
* Women of child-bearing potential* must have a negative pregnancy test in serum or urine before the inclusion in the study and agree to use highly effective contraceptive methods during the study. Highly effective contraceptive methods will include: intrauterine device, bilateral tubal occlusion, vasectomized partner and sexual abstinence.
* Hormonal contraceptive methods will be avoided due to the risk of adverse events and impairment of liver function.

Exclusion Criteria:

* Presence of other respiratory disorders, (i.e. current physician diagnosis of asthma, early life history of asthma (<21 years) a previous clinical diagnosis of bronchiectasis, interstitial lung disease, pulmonary eosinophilia).
* Long-term oxygen therapy or non-invasive mechanical ventilation at home.
* Current smokers.
* Active cancer.
* Use of ICS in the 3 months prior to the recruitment.
* Participating in another randomized trial.
* Not likely to complete the study.
* Pregnant or breastfeeding females.
* Exacerbations in the previous 8 weeks.
* Primary or secondary immunodeficiency.
* Immunosuppression or regular oral corticosteroid treatment.
* Allergy to IMP's excipients.
* Any circumstances which could contradict study participation and lead the investigator to assess the patient as unsuitable for study participation for any other reason.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Significant molecular changes in COPD stratified by their blood eosinophil counts. | 8 weeks
  Significant molecular changes (p<0.05, and/or FDR<0.05) (e.g. microbiome and/or transcriptome and/or proteins and/or epigenetics) in sputum, nasal and oropharyngeal swabs, urine and/or blood associated with ICS treatment vs. no ICS treatment (usual care), in COPD stratified by their blood eosinophil counts.

SECONDARY OUTCOMES:
Significant molecular changes in COPD with different airflow limitation severities. | 8 weeks
  Significant molecular changes (p<0.05, and/or FDR<0.05) (e.g. microbiome and/or transcriptome and/or proteins and/or epigenetics) in sputum, nasal and oropharyngeal swabs, urine and/or blood associated with ICS treatment vs. no ICS treatment (usual care), in COPD with different airflow limitation severities.

CONTACTS AND LOCATIONS:
Locations (6):
- Philips University of Marburg, Marburg, Germany
- Academisch Ziekenhuis Groningen, Groningen, Netherlands
- Spain (2):
  - Clínic Barcelona, Barcelona
  - Son Espases, Palma de Mallorca
- United Kingdom (2):
  - University of Leicester, Leicester
  - Imperial College London, London